CLINICAL TRIAL: NCT00884091
Title: A Pilot Study to Evaluate the Glucagon-Like Peptide 1 Response to the Challenge of Mixed Meals in Chinese Subjects
Acronym: IC-1-V1
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Attending physician, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 98-01-48A
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: Chinese; Glucagon-like peptide 1; Glucagon; Insulin; Mixed meals; Healthy Adults
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma samples retained, with no potential for DNA extraction from any retained samples. The retained samples will be destroyed after the results published.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Adults: 1. Chinese in origin
  2. Healthy
  3. No medication at least two weeks before the study

SUMMARY:
The purpose of the study is to standardize a meal test to facilitate future studies of the postprandial glucagons-like peptide 1 (GLP-1) response in Chinese subjects. Eighteen healthy Chinese subjects, aged between 20-65 years old, without history of diabetes, will be recruited for the study. Each subject will receive two mixed meal tests for postprandial GLP-1 excursion at random order: 60 % carbohydrate (CHO)/20 % fat vs. 50 % CHO/30 % fat. The postprandial glucose, insulin, glucagon and other related hormones responses will also be measured. Through the study, we hope to build up a platform for the study of the postprandial GLP-1 response and insulin secretion.

DETAILED DESCRIPTION:
Glucagon-like peptide 1 (GLP-1) is a 30-amino acid peptide produced in the intestinal epithelial endocrine L-cells. It stimulates insulin and suppresses glucagons secretion, inhibits gastric emptying, and reduces appetite and food intake. In the fasting state, the plasma concentrations of GLP-1 are very low. Levels of circulating GLP-1 rise rapidly after food intake. The GLP-1 meal response depends on ingested nutrients. Carbohydrates are strong stimuli of GLP-1 release. Protein stimulates GLP-1 release, even more than carbohydrates. GLP-1 concentrations also increase after intake of fat, although the elevation is delayed compared to the stimulation of carbohydrates. Dietary fibers may also modify the postprandial GLP-1 response. Therefore, it is essential for us to characterize nutrient compositions of test meals for further studies of meal response of GLP-1.

Other sampling conditions of the meal tests are also needed to be taking care of. GLP-1 is rapidly degraded by the enzyme dipeptidyl peptidase IV (DPP-4). During the meal tests, it is important adding enzyme inhibitors into sampling tubes to avoid hormone degradation. Lugari et al. collected blood samples into tubes containing EDTA and aprotinin during a meal test. They could obtain samples from the same tube for both glucagons and GLP-1 assays. Other study groups reported that samples for GLP-1 needed to be collected into Vacutainer tubes prepared with EDTA and DPP-4 inhibitor for preventing degradation of GLP-1. Another aim of the present study is to compare the differences in GLP-1 concentrations in samples collected by EDTA tubes containing aprotinin or a DPP-4 inhibitor during the meal tests.

Racial differences in GLP-1 levels during oral glucose challenge have been demonstrated recently that severely obese African Americans exhibited lower GLP-1 concentrations than Caucasians. It is worthwhile to examine the meal response of GLP-1 across ethnicities. The current study proposes to observe the GLP-1 response during standardized meal tests in a group of Chinese subjects.

The purpose of the study is to standardize a meal test to facilitate future studies of the postprandial GLP-1 response in Chinese subjects. Eighteen healthy Chinese subjects, aged between 20-65 years old, without history of diabetes, will be recruited for the study. Each subject will receive two mixed meal tests for postprandial GLP-1 excursion at random order: 60 % carbohydrate (CHO)/20 % fat vs. 50 % CHO/30 % fat. The postprandial glucose, insulin, glucagon and other related hormones responses will also be measured. Through the study, we hope to build up a platform for the study of the postprandial GLP-1 response and insulin secretion.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 20 ~ 65 years old.
* Willing to participate by signing an informed consent.
* Willing to undergo two standardized mixed meal test at two separate visits

Exclusion Criteria:

* Patients of known history of type 2 diabetes.
* History of major renal, liver, heart, blood and neurological disease.
* History of alcoholism or drug abuse.
* Women who are pregnant.
* Current or concomitant illness that would interfere with the subject's ability to perform the study or that would confound the study results, judged by the investigation physicians.
* Any concomitant medication within 2 weeks of the study.
* Difficult venous access

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Invited normal healthy volunteers from a research clinic
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
the differences in post-challenge GLP-1 responses between the two meal tests | 8 months

SECONDARY OUTCOMES:
the correlations of incremental GLP-1 response with insulin sensitivity and insulin secretion indices in each of the meal test | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Min Hwu, MD, Principal Investigator — Taipei Veterans eneral Hospital
Locations (1):
- Section of Endocrinology and Metabolism, Department of Medicine, Taipei Veterans General Hospital, Taipei, Taiwan